CLINICAL TRIAL: NCT06730022
Title: Dermacyte® Liquid for Treatment of Cutaneous Ulcers and Wounds
Status: Available | Type: Expanded Access
Sponsor: Merakris Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: DL-EAP-201
Record Dates: First submitted 2024-12-06; First posted 2024-12-12 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cutaneous Ulcer; Diabetic Ulcer; Surgical Wound Dehiscence; Burns - Multiple; Pressure Ulcers; Mixed Ulcer; Ischemic Ulcer
MeSH Terms: conditions — Skin Ulcer; Surgical Wound Dehiscence; Pressure Ulcer

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: MTX-001 (Dermacyte Liquid) — Repeat dose subcutaneous drug injection for the treatment of serious chronic wounds.

SUMMARY:
The objective of this study is to make Dermacyte Liquid available on an expanded access basis to treat cutaneous ulcers and wounds refractory to initial treatment or that do not have adequate alternative treatments. Minimal data will be collected to evaluate the efficacy and safety of Dermacyte Liquid.

DETAILED DESCRIPTION:
The primary purpose is to provide expanded access of Dermacyte Liquid to subjects who have serious cutaneous ulcers and wounds (e.g., ulcers related to diabetes mellitus, venous insufficiency, complications of systemic sclerosis or rheumatic disease; decubitus ulcers, burns, acute trauma, wound dehiscence, ischemic ulcers, and mixed etiology ulcers). Eligible subjects must have a high likelihood of significant morbidity, loss of quality of life, potential amputation, or mortality without efficacious treatment. As there are many types of patients who may be enrolled, study results will not have statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Must have a cutaneous ulcer or wound refractory to initial treatment or does not have an adequate treatment alternative, as determined by the Investigator

Exclusion Criteria:

* Must not be pregnant or lactating
* Must not have known malignancies
* Must not be less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- The WISH Clinic, Arvada, Colorado, United States